CLINICAL TRIAL: NCT03502239
Title: Cognitive Rehabilitation (Mega Team) and Its Effects on Emotional and Behavioral Regulation in ADHD, ASD, and CHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Child-Bright Network (Other); Ehave (Other); The Governors of the University of Alberta (Unknown)
Responsible Party: Principal Investigator, Jennifer Crosbie, Clinical Scientist/Psychologist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1000057380
Record Dates: First submitted 2018-03-12; First posted 2018-04-18 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: ADHD; ASD; CHD - Congenital Heart Disease
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Heart Defects, Congenital

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group (Experimental): Subjects randomly assigned to this arm will train on the Mega Team video game.
  Interventions: Other: Mega Team - video game
- Control- wait list group (No Intervention): Subjects randomly assigned to this arm will be the wait-list group. They are allowed to play the video games that they usually play.

INTERVENTIONS:
Other: Mega Team - video game — Subjects randomly assigned to the treatment group will be instructed to practice Mega Team for 15 minutes a day, 5 days a week for a minimum of 21 days and a maximum of 25 days.
  Other Names: Mega Team
  Arms: Treatment group

SUMMARY:
Children with disorders that impact neurodevelopment often have difficulties with executive functions and regulating emotions. Cognitive-based video game training has been shown to improve outcomes, however, this training has been expensive, has required professional supervision, and has been investigated only within a narrow group of children. The Mega Team study will test the effects of a highly engaging, take-home video game-based intervention designed to improve executive functioning in children with various brain-based developmental disorders.

DETAILED DESCRIPTION:
The target population for this study will be children between the ages of 6-12 with a diagnosis of ADHD, ASD or CHD. Potential subjects for this study will be recruited from the clinical teams within SickKids and partnering institutions (e.g., CAMH and Holland Bloorview). Participants will be identified by a psychiatrist, psychologist or specialist physician as meeting diagnostic criteria for one of the three disorders; 1) ADHD, 2) ASD, 3) CHD. Families of children who have expressed interested in this study will be contacted by research staff to discuss the study in more detail and will coordinate the logistics of an initial consent and enrollment appointment. Parent(s)/guardian(s) of participants will be required to consent and children will be required to assent to take in this study.

This protocol is divided into 3 studies: sub-study 1 (ADHD), sub-study 2 (ASD) and sub-study 3 (CHD) each consisting of a pre-post treatment design with 6 month follow-up. Each sub-study includes an active treatment and wait -list arm. Please see study visit schedule (pg. 11) for time-line of events and measures by participant at each time point. Participants will be tested at SickKids at pre-treatment, post-treatment and follow-up. Participants will train at home with weekly calls from research staff. Assessors at all clinic visits will be blind to treatment status. All pre, post and following-up clinic assessments will be conducted off stimulant medication with a washout period of 48 hours.

Stratification: Participants may be taking medications at the time of the study (stimulants and non-stimulants including SSRI or antipsychotic medications). Families will be asked to be stabilized on their current dose of medication for at least for a month before commencing the study and to maintain the same medication and dosage during the 5 week study. If a change in the type of medication or dosage takes place during the study it will be recorded. Due to the established impact of stimulant medications on EF 20 21 this class of medication will be used as part of the randomization process to attain equal proportions of participants using stimulant medications in the Mega Team and TAU groups. As some medication use is anticipated in all disorder groups the same randomization approach will be used in all three studies.

Sample Size: The sample size for sub-study 1 (ADHD) will be 220 participants with 110 randomized into each group from initial estimated recruitment pool of 250. The sample size will provide 80% power to declare statistical significance if the true difference between treatment groups is 0.43 standard deviations or greater, using a two-sided, 5% level test of hypothesis, Bonferroni corrected for three comparisons. A pilot study of Mega Team is currently underway (Dr. Crosbie PI, a registered clinical trial) and results from that pilot will provide final estimates of the standard deviations before commencement of the current study. The planned sample for each of sub-study 2 (ASD) and sub-study 3 (CHD) will be 120 (60 per arm) given the novelty of investigating cognitive rehabilitation targeting EFs in these populations. Information from sub-study 1, which will happen first, and the results from the Mega Team pilot study, will allow adjustment in sample size of sub-study 2 and sub-study 3. All aspects of enrollment, randomization, and attrition will be monitored and documents using CONSORT flow diagram22.

Randomization: Participants within each sub-study who have consented/ assented to the study and meet all inclusion criterion will be randomized to either Mega Team or TAU waitlist stratified by medication status (yes or no)) using random block sizes. Randomization will be carried out using RedCAP23.

Blinding: Assessors at all clinic visits will be blind to treatment status. Participants and parents will be asked not to make mention of their treatment status during visits. They will be reminded of this regularly. Assessors will indicate their blinded status at the end of all visits. Parents and children will be asked not to inform teachers of the treatment status. At the time of questionnaire completion, teachers will be asked if they are aware of the treatment status of the child.

Intervention Conditions:

Mega Team Training Sessions: Mega Team is highly engaging video game based cognitive intervention that trains multiple executive functions: response inhibition, verbal working memory and visual working memory in the context of a single game with increasing difficulty based on the individual performance. Children in the treatment group will train at home on their own tablet or on a study tablet provided to the family (if needed). They will be instructed to practice Mega Team for 15 minutes a day, approximately 5 days a week for a targeted minimum of 21 sessions and a maximum of 25 sessions. The minimum value of 21 sessions has been selected based on findings of prior research. Majority of studies using other models of intervention have been able to capture significant training-induced improvements after 21 sessions 24-26. The maximum training of 25 sessions has been set to control for variability within and between our groups. Performance on Mega Team will automatically upload to a secure portal hosted by eHave for monitoring of enrolment, adherence and for data analyses. Scoring algorithms will track how often and how long the participants trained on Mega Team as well as their performance. Weekly calls from research staff will provide motivation and address barriers to game play.

TAU waiting list Control: Children in the control group will not be provided with any overt intervention but continue with treatment recommendations as provided by their clinical care team. They will be asked to complete a video game usage log weekly to record the type and duration of their regular video game playing, and will receive weekly calls from research staff, as will participants assigned to Mega Team. Participants on in the TAU group will be given access to the game at the completion of the 6 month follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Sub-Study 1 Inclusion Criteria

  1. Must be 6-12 years of age
  2. Have IQ above 70 as estimated by two subtests of the Wechsler Abbreviated Scale of intelligence, Second Edition (WASI II) or equivalent.
  3. Diagnosed with ADHD based upon DSM 5 criteria by a referring clinician confirmed by semi structured interview with the parents using PICS, including information from parent and teacher ratings of an established measure of ADHD symptoms.
  4. Does not have a diagnosis of ASD or CHD [in this case, individuals can be enrolled into Study 2 (ASD) or Study 3 (CHD)].
  5. Have reliable access to the internet
* Sub-Study 2 inclusion criteria

  1. Must be 6-12 years of age
  2. Have IQ above 70 as estimated by two subtests of the Wechsler Abbreviated Scale of intelligence, Second Edition (WASI II) or equivalent
  3. Meets clinical diagnosis of ASD by referral services (Holland Bloorview, CAMH) supported by ADOS.
  4. Have reliable access to the internet
* Sub-Study 3 inclusion criteria

  1. Must be 6-12 years of age
  2. Have IQ above 70 as estimated by two subtests of the Wechsler Abbreviated Scale of intelligence, Second Edition (WASI II) or equivalent
  3. Must have a diagnosis of Transposition of the Great Arteries (TGA) or Hypoplastic left heart syndrome
  4. Must have received cardiac surgery before 6 weeks of age.
  5. Have reliable access to the internet

Exclusion Criteria:

* Sub-Study 1 Exclusion Criteria

  1. Younger than 6 years or older than 12
  2. IQ below 70 as estimated by two subtests of the Wechsler Abbreviated Scale of intelligence, Second Edition (WASI II) or equivalent
  3. Does not meet consensus diagnosis of DSM 5 criteria for ADHD based on a semi structured interview with the parents using PICS-6, including information from parent and teacher ratings of an established measure of ADHD symptoms.
  4. Has a diagnosis of ASD or CHD [in this case, individuals can be enrolled into Study 2 (ASD) or Study 3 (CHD)].
* Sub-Study 2 exclusion criteria

  1. Younger than 6 years or older than 12
  2. IQ below 70 as estimated by two subtests of the Wechsler Abbreviated Scale of intelligence, Second Edition (WASI II) or equivalent
  3. Does not meet confirmed diagnosis of ASD based on ADOS
* Sub-Study 3 exclusion criteria

  1. Younger than 6 years or older than 12
  2. IQ below 70 as estimated by two subtests of the Wechsler Abbreviated Scale of intelligence, Second Edition (WASI II) or equivalent
  3. Does not have a diagnosis of Transposition of the Great Arteries (TGA) or Hypoplastic left heart syndrome
  4. Did not receive cardiac surgery before 6 weeks of age.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 440 (Actual)
Dates: Start 2018-05-26 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Change in Response Inhibition | Baseline, Post-training study visit #1 (4-5 weeks after baseline), Post-training study visit #2 (6 months after baseline)
  Inhibitory control will be measured using the Stop Signal Task (SST). The SST measures the ability to cancel an already initiated motor response. The primary outcome measure will be the participants' average stop signal reaction time (SSRT).
Change in Working Memory | Baseline, Post-training study visit #1 (4-5 weeks after baseline), Post-training study visit #2 (6 months after baseline)
  Verbal and Spatial N-back (1, 2 conditions) will be used to assess central executive working memory. The N-Back task requires on-line monitoring, updating, and manipulation of information and measures key processes within working memory. In the N-Back task, the participant is required to monitor a series of stimuli and to respond whenever a stimulus is presented that is the same as the one presented n trials previously, where n is a pre-specified integer, usually 0, 1, or 2. The current study will use letters (verbal) and spatial location (spatial) paradigms. Visual and spatial working memory span will be assessed using the Spatial Span subtest and the Digit Span item from the WISC-IV Integrated. The primary outcome measure will be the overall score.

SECONDARY OUTCOMES:
Planning and Organization | Baseline, Post-training study visit #1 (4-5 weeks after baseline), Post-training study visit #2 (6 months after baseline)
  The Tower Test from the Delis-Kaplan Executive Function System (D-KEFS;28 is a test of planning and problem solving abilities. Participants are asked to construct towers of discs on a set of pegs corresponding to a model. Raw scores reflect the participant's ability to use the fewest possible moves to achieve the tower depicted in the model.
Everyday functioning and impairment | Baseline, Post-training study visit #1 (4-5 weeks after baseline), Post-training study visit #2 (6 months after baseline)
  Parent and teacher rating of behaviours and impairments associated with executive functions will be assessed using The Behavior Rating Inventory of Executive Function (BRIEF;29). This is a 86 item questionnaires with solid psychometric properties (ref) with correlations with other measures of emotional and behavioral functioning29.
Inattentive and Hyperactivity Behaviour rated by parent and teacher | Baseline, Post-training study visit #1 (4-5 weeks after baseline), Post-training study visit #2 (6 months after baseline)
  Items associated with inattentiveness and hyperactivity from the SNAP IV will be used to estimate behavioural symptoms associated with ADHD. The SNAP-IV (SNAP-IV; Swanson IV, 2003) is an 18-item scale that includes the DSM-IV criteria for ADHD with items 1-9 representing the inattentive subset of symptoms and items 10-18 representing the Hyperactivity/Impulsivity subset.
Academic accuracy and efficiency | Baseline, Post-training study visit #1 (4-5 weeks after baseline), Post-training study visit #2 (6 months after baseline)
  Academic efficiency and accuracy will be assessed using the fluency measures from the Woodcock Johnson III30 test of achievement. The fluency tasks measure the accuracy of completing academic tasks within a time limit. Reading, math and writing fluency subtests will be included.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Crosbie, Ph.D., C.Psych., Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
de-identified data will be shared with our sponsor/funders - ChildBright Network and eHave.

REFERENCES:
- [Background] Diamond A. Executive functions. Annu Rev Psychol. 2013;64:135-68. doi: 10.1146/annurev-psych-113011-143750. Epub 2012 Sep 27. PMID 23020641
- [Background] McAuley T, Crosbie J, Charach A, Schachar R. The persistence of cognitive deficits in remitted and unremitted ADHD: a case for the state-independence of response inhibition. J Child Psychol Psychiatry. 2014 Mar;55(3):292-300. doi: 10.1111/jcpp.12160. Epub 2013 Nov 22. PMID 24261515
- [Background] Lawson RA, Papadakis AA, Higginson CI, Barnett JE, Wills MC, Strang JF, Wallace GL, Kenworthy L. Everyday executive function impairments predict comorbid psychopathology in autism spectrum and attention deficit hyperactivity disorders. Neuropsychology. 2015 May;29(3):445-53. doi: 10.1037/neu0000145. Epub 2014 Oct 13. PMID 25313979
- [Background] Morris MC, Evans LD, Rao U, Garber J. Executive function moderates the relation between coping and depressive symptoms. Anxiety Stress Coping. 2015;28(1):31-49. doi: 10.1080/10615806.2014.925545. Epub 2014 Jun 17. PMID 24866556
- [Background] Vinogradov S, Fisher M, de Villers-Sidani E. Cognitive training for impaired neural systems in neuropsychiatric illness. Neuropsychopharmacology. 2012 Jan;37(1):43-76. doi: 10.1038/npp.2011.251. Epub 2011 Nov 2. PMID 22048465
- [Background] Cortese S, Ferrin M, Brandeis D, Buitelaar J, Daley D, Dittmann RW, Holtmann M, Santosh P, Stevenson J, Stringaris A, Zuddas A, Sonuga-Barke EJ; European ADHD Guidelines Group (EAGG). Cognitive training for attention-deficit/hyperactivity disorder: meta-analysis of clinical and neuropsychological outcomes from randomized controlled trials. J Am Acad Child Adolesc Psychiatry. 2015 Mar;54(3):164-74. doi: 10.1016/j.jaac.2014.12.010. Epub 2014 Dec 29. PMID 25721181
- [Background] Beck SJ, Hanson CA, Puffenberger SS, Benninger KL, Benninger WB. A controlled trial of working memory training for children and adolescents with ADHD. J Clin Child Adolesc Psychol. 2010;39(6):825-36. doi: 10.1080/15374416.2010.517162. PMID 21058129
- [Background] Dahlin, K. I. E. Effects of working memory training on reading in children with special needs. Read. Writ. 24, 479-491 (2011)
- [Background] Holmes J, Gathercole SE, Dunning DL. Adaptive training leads to sustained enhancement of poor working memory in children. Dev Sci. 2009 Jul;12(4):F9-15. doi: 10.1111/j.1467-7687.2009.00848.x. PMID 19635074
- [Background] Johnstone SJ, Roodenrys S, Blackman R, Johnston E, Loveday K, Mantz S, Barratt MF. Neurocognitive training for children with and without AD/HD. Atten Defic Hyperact Disord. 2012 Mar;4(1):11-23. doi: 10.1007/s12402-011-0069-8. Epub 2011 Dec 20. PMID 22179720
- [Background] Alloway, T. Can interactive working memory training improving learning? J. Interact. Learn. Res. 23, 197-207 (2012)
- [Background] Shalev L, Tsal Y, Mevorach C. Computerized progressive attentional training (CPAT) program: effective direct intervention for children with ADHD. Child Neuropsychol. 2007 Jul;13(4):382-8. doi: 10.1080/09297040600770787. PMID 17564853
- [Background] Van der Molen MJ, Van Luit JE, Van der Molen MW, Jongmans MJ. Everyday memory and working memory in adolescents with mild intellectual disability. Am J Intellect Dev Disabil. 2010 May;115(3):207-17. doi: 10.1352/1944-7558-115.3.207. PMID 20441391
- [Background] Craig F, Margari F, Legrottaglie AR, Palumbi R, de Giambattista C, Margari L. A review of executive function deficits in autism spectrum disorder and attention-deficit/hyperactivity disorder. Neuropsychiatr Dis Treat. 2016 May 12;12:1191-202. doi: 10.2147/NDT.S104620. eCollection 2016. PMID 27274255
- [Background] Willcutt EG, Doyle AE, Nigg JT, Faraone SV, Pennington BF. Validity of the executive function theory of attention-deficit/hyperactivity disorder: a meta-analytic review. Biol Psychiatry. 2005 Jun 1;57(11):1336-46. doi: 10.1016/j.biopsych.2005.02.006. PMID 15950006
- [Background] Calderon J, Bellinger DC. Executive function deficits in congenital heart disease: why is intervention important? Cardiol Young. 2015 Oct;25(7):1238-46. doi: 10.1017/S1047951115001134. Epub 2015 Jun 17. PMID 26082199
- [Background] Wechsler, D. WASI -II: Wechsler abbreviated scale of intelligence - second edition. J. Psychoeduc. Assess. 31, 337-41 (2013)
- [Background] Kaufman J, Birmaher B, Brent D, Rao U, Flynn C, Moreci P, Williamson D, Ryan N. Schedule for Affective Disorders and Schizophrenia for School-Age Children-Present and Lifetime Version (K-SADS-PL): initial reliability and validity data. J Am Acad Child Adolesc Psychiatry. 1997 Jul;36(7):980-8. doi: 10.1097/00004583-199707000-00021. PMID 9204677
- [Background] Bussing R, Fernandez M, Harwood M, Wei Hou, Garvan CW, Eyberg SM, Swanson JM. Parent and teacher SNAP-IV ratings of attention deficit hyperactivity disorder symptoms: psychometric properties and normative ratings from a school district sample. Assessment. 2008 Sep;15(3):317-28. doi: 10.1177/1073191107313888. Epub 2008 Feb 29. PMID 18310593
- [Background] Bedard AC, Ickowicz A, Logan GD, Hogg-Johnson S, Schachar R, Tannock R. Selective inhibition in children with attention-deficit hyperactivity disorder off and on stimulant medication. J Abnorm Child Psychol. 2003 Jun;31(3):315-27. doi: 10.1023/a:1023285614844. PMID 12774864
- [Background] Bedard AC, Martinussen R, Ickowicz A, Tannock R. Methylphenidate improves visual-spatial memory in children with attention-deficit/hyperactivity disorder. J Am Acad Child Adolesc Psychiatry. 2004 Mar;43(3):260-8. doi: 10.1097/00004583-200403000-00006. PMID 15076258
- [Background] Boutron I, Moher D, Altman DG, Schulz KF, Ravaud P; CONSORT Group. Extending the CONSORT statement to randomized trials of nonpharmacologic treatment: explanation and elaboration. Ann Intern Med. 2008 Feb 19;148(4):295-309. doi: 10.7326/0003-4819-148-4-200802190-00008. PMID 18283207
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Chein JM, Morrison AB. Expanding the mind's workspace: training and transfer effects with a complex working memory span task. Psychon Bull Rev. 2010 Apr;17(2):193-9. doi: 10.3758/PBR.17.2.193. PMID 20382919
- [Background] Dahlin E, Nyberg L, Backman L, Neely AS. Plasticity of executive functioning in young and older adults: immediate training gains, transfer, and long-term maintenance. Psychol Aging. 2008 Dec;23(4):720-30. doi: 10.1037/a0014296. PMID 19140643
- [Background] Jaeggi SM, Buschkuehl M, Jonides J, Perrig WJ. Improving fluid intelligence with training on working memory. Proc Natl Acad Sci U S A. 2008 May 13;105(19):6829-33. doi: 10.1073/pnas.0801268105. Epub 2008 Apr 28. PMID 18443283
- [Background] Logan, G. D., Schachar, R. J. & Tannock, R. Impulsivity and Inhibitory Control. Psychol. Sci. 8, 60-64 (1997)
- [Background] Delis, D., Kaplan, E. & Kramer, J. Delis-Kaplan executive function system (D-KEFS). Can. J. Sch. Psychol. 20, 117-128 (2001)
- [Background] Baron IS. Behavior rating inventory of executive function. Child Neuropsychol. 2000 Sep;6(3):235-8. doi: 10.1076/chin.6.3.235.3152. No abstract available. PMID 11419452
- [Background] Woodcock, R. W., McGrew, K. S. & Mather, N. Woodcock-Johnson III Tests of Achievement. Test 2001, 1-9 (2001)